CLINICAL TRIAL: NCT06704074
Title: Effectiveness of Real Home Settings Via Virtual Reality Task Oriented Training on Upper Limb Function in Patients With Stroke
Brief Title: Virtual Reality Task Oriented Training on Upper Limb Function in Stroke Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Collaborators: First Affiliated Hospital of Chongqing Medical University (Other); Shanghai Yangzhi Rehabilitation Hospital (Unknown); Beihang University (Other); Huashan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KYLL-202408-001-1
Record Dates: First submitted 2024-11-11; First posted 2024-11-25 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Stroke
Keywords: stroke; rehabilitation; Task-oriented training (TOT); virtual reality (VR); upper limb dysfunction
MeSH Terms: conditions — Stroke | interventions — Smart Glasses

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- VR+TOT (task oriented training combined with occupational training) (Experimental): The participants in this group are given VR-TOT training, which was created a virtual scene based on the participants' home and completed a series of occupational tasks. A Head-mounted-display VR device is used in this group.
  Interventions: Device: virtual reality (VR) head mounted display
- TOT (task oriented training) (Other): In this group, the occupational task is selected according to the level of the upper limb function assessment , and all the training programs are related to the activities of daily life (ADL).
  Interventions: Device: virtual reality (VR) head mounted display
- Traditional OT (No Intervention): Traditional OT , including but not limited : upper limb joints (shoulder, elbow, wrist, interphalangeal), muscle sensory stimulation (such as tapping, brushing, squeezing, etc.), active and passive range of motion training of upper limb joints, upper limb muscle strength training, wrist dorsal extension, grip and other training were carried out by using a roller and wooden nail board. ADL training (dressing, grooming, washing, eating, etc.).

INTERVENTIONS:
Device: virtual reality (VR) head mounted display — The participants' in this group were given VR-TOT training under real home scenes created in the platform of Unity. There were 6 VR-TOT tasks, and the task choice was according to the performance of participants' upper limb function. The experienced therapist will guide and monitor the participants and adjust the task if necessary.
  Arms: TOT (task oriented training); VR+TOT (task oriented training combined with occupational training)

SUMMARY:
Stroke rank second among the top causes of death, affecting millions of people in the worldwide. It has been reported that hemiplegia is the most common sequelae after stroke, accounting for about 50%-70% of all sequelae of the disease. About 75% of stroke patients are accompanied by different degrees of upper limb dysfunction, which seriously affects the activities of daily life and cause serious physical and mental burden to patients and their families. Early recovery of upper limb motor function is a great significance for the overall recovery of stroke patients. Task-oriented training (TOT) is reported to improve the motor coordination and ADL. However, lack varies of tasks limited the treatment ability for patients with stroke hemiplegia during hospital admission. Virtual reality (VR) offers advantages of providing virtual scenes that is difficult in the real world, such as the scene of garden, camara, and plaza etc. And the familiar circumstances for patients may have the potential to increase the motivation of rehabilitation training, and improve the efficacy of occupational therapy (OT).

The goal of this study is to observe the effectiveness of real home settings via virtual reality assisted TOT on upper limb function in patients with stroke. Functional near-infrared spectroscopy (fNIRS) and electroencephalography (EEG) were used to observe the changes in brain function under VR-TOT training.

We intended to recruit 120 participants, and allocate to three groups: VR-TOT, TOT, and traditional OT. Each of them completed the Fugl-Meyer-UE, Wolf motor function test (WMFT), hand gripping power, modified Ashworth、Purdue Pegboard test （PPT）、modified Barthel index (MBI)、mini mental state examination (MMSE)、NIH stroke scale (NIHSS)、Virtual reality sickness questionnaire (VRSQ), Intrinsic Motivation Inventory Inventory (IMI), satisfaction VAS, body representation, sense of ownership, Proprioceptive Drift scale before and after the treatment. Additionally, we conducted fNIRS and EEG at baseline and during the follow up to understand the changes in brain function.

ELIGIBILITY:
Inclusion Criteria:

-1. Ischemic or hemorrhagic stroke was diagnosed based on the history, symptoms, and signs combined with CT or MRI imaging; 2. First stroke, onset time from 1 to 6 months, age ≥ 18 - 80 years ; 3. Hemiplegia, Brunnstrom stage > Ⅰ, modified Ashworth grade < 4; 4. Patients can sit and stand for upper limb function assessment and rehabilitation training; 5. No severe cognitive impairment, MMSE > 17, able to accurately understand the questionnaire questions and scoring criteria, and complete the body drift test; No history of serious mental illness; 6. No obvious abnormality in visual acuity or corrected visual acuity; There was no obvious abnormality in hearing. There was no sensory aphasia or unilateral neglect.

7. Patients or their family members signed informed consent to participate in the experiment.

Exclusion Criteria:

* 1. Previous history of stroke, traumatic or non-vascular encephalopathy; 2. Skull defect or allogeneic repair; 3. combined with other neurological and mental diseases; 4. Previous diseases that may cause upper limb motor/sensory dysfunction, such as neck tumor or radiotherapy and chemotherapy history, cervical spondylosis, cervical spine or upper limb fracture history, traumatic brachial plexus injury history, arthritis, diabetes mellitus, myasthenia gravis, multiple sclerosis, etc.

  5. Accompanied by obvious vertigo or dizziness symptoms or related diseases (such as motion sickness, Meniere's syndrome, otolithiasis, etc.); 6. Accompanied by obvious pain; 7. Evidence of ataxia and cerebellar or brainstem lesions according to the NIHSS; 8. Ongoing participation in other clinical investigators; 9. Unstable condition, refusal to sign the informed consent, and unwillingness to cooperate with the examination and treatment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 120 (Estimated)
Dates: Start 2025-03-09 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment Upper Extremity Scale (FAM-UE) | There were 3 time points for evaluation:after screening for enrollment but before study initiation,the intervention of 2 weeks, the intervention of 4 weeks

SECONDARY OUTCOMES:
Wolf motor function test（WMFT） | There were 3 time points for evaluation:after screening for enrollment but before study initiation,the intervention of 2 weeks, the intervention of 4 weeks
The grip strength of the hand | There were 3 time points for evaluation:after screening for enrollment but before study initiation,the intervention of 2 weeks, the intervention of 4 weeks
the Modified Ashworth scale | There were 3 time points for evaluation:after screening for enrollment but before study initiation,the intervention of 2 weeks, the intervention of 4 weeks
Box and Block Test（BBT） | There were 3 time points for evaluation:after screening for enrollment but before study initiation,the intervention of 2 weeks, the intervention of 4 weeks
Modified Barthel Index Scale(MBI) | There were 3 time points for evaluation:after screening for enrollment but before study initiation,the intervention of 2 weeks, the intervention of 4 weeks
Intrinsci Motivation Inventory (IMI) | There were 3 time points for evaluation: after screening for enrollment but before study initiation, the intervention of 2 weeks, the intervention of 4 weeks
Visual Analogue Scale（VAS） | the intervention of 2 weeks, the intervention of 4 weeks
the sense of ownership (SOO) | There were 3 time points for evaluation:after screening for enrollment but before study initiation,the intervention of 2 weeks, the intervention of 4 weeks
the questionnaire and self-location drift | There were 3 time points for evaluation: after screening for enrollment but before study initiation, the intervention of 2 weeks, the intervention of 4 weeks
fNIRS | There were 3 time points for evaluation: after screening for enrollment but before study initiation, the intervention of 2 weeks, the intervention of 4 weeks
EEG | There were 3 time points for evaluation: after screening for enrollment but before study initiation, the intervention of 2 weeks, the intervention of 4 weeks
Catherine Bergego Scale（CBS） | There were 3 time points for evaluation:after screening for enrollment but before study initiation,the intervention of 2 weeks, the intervention of 4 weeks
line bisection test | There were 3 time points for evaluation:after screening for enrollment but before study initiation,the intervention of 2 weeks, the intervention of 4 weeks

OTHER OUTCOMES:
Mini Mental State Examination(MMSE) | screening for enrollment
National Institute of Health Stroke Scale(NIHSS) | after screening for enrollment but before study initiation
the Virtual Reality Symptom Questionnaire(VRSQ) | the intervention of 2 weeks, the intervention of 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- a Head-mounted-display VR device, Jinan, Shangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Malik AN, Masood T. Task-oriented training and exer-gaming for improving mobility after stroke: A randomized trial. J Pak Med Assoc. 2021 Jan;71(1(B)):186-190. doi: 10.47391/JPMA.560. PMID 35157646
- [Background] Jeong S, Chung Y. Task-Oriented Training with Abdominal Drawing-in Maneuver in Sitting Position for Trunk Control, Balance, and Activities of Daily Living in Patients with Stroke: A Pilot Randomized Controlled Trial. Healthcare (Basel). 2023 Dec 4;11(23):3092. doi: 10.3390/healthcare11233092. PMID 38063660
- [Background] Cano-de-la-Cuerda R. Influential Women in the Field of Neurological Rehabilitation: A Literature Review. Int J Environ Res Public Health. 2022 Jan 20;19(3):1112. doi: 10.3390/ijerph19031112. PMID 35162136
- [Background] Huang J, Ji JR, Liang C, Zhang YZ, Sun HC, Yan YH, Xing XB. Effects of physical therapy-based rehabilitation on recovery of upper limb motor function after stroke in adults: a systematic review and meta-analysis of randomized controlled trials. Ann Palliat Med. 2022 Feb;11(2):521-531. doi: 10.21037/apm-21-3710. PMID 35249330
- See also: The Effect of Task-Oriented Activities Training on Upper-Limb Function, Daily Activities, and Quality of Life in Chronic Stroke Patients: A Randomized Controlled Trial — https://pubmed.ncbi.nlm.nih.gov/36361001/
- See also: Effects of task-oriented training on upper extremity function and performance of daily activities by chronic stroke patients — https://pubmed.ncbi.nlm.nih.gov/26355425/
- See also: task-oriented training in the treatment of developmental coordination disorder — http://www.cjpmr.cn/ch/reader/create_pdf.aspx?file_no=2023030284&flag=1&journal_id=zhwlyxykf&year_id=2023
- See also: observe the effect of a family-centered task-oriented training (TOT) program on the functional independence and life quality of children with spastic cerebral palsy — http://www.cjpmr.cn/ch/reader/create_pdf.aspx?file_no=2022020138&flag=1&journal_id=zhwlyxykf&year_id=2022
- See also: observe any effect of task-oriented training in the activities of daily living (ADL) for stroke patients. — http://www.cjpmr.cn/ch/reader/view_abstract.aspx?file_no=2022070595&flag=1